CLINICAL TRIAL: NCT06858228
Title: Comparison of Denervation Techniques for the Treatment of Knee Osteoarthritis: a Randomized Clinical Trial of Continuous Ablative Radiofrequency Vs. Chemical Denervation with Absolute Alcohol
Brief Title: Comparison of Denervation Techniques for the Treatment of Knee Osteoarthritis: Continuous Ablative Radiofrequency Vs. Chemical Denervation with Absolute Alcohol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Henrique Cunha Ferraro, Associate Professor, MD, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 85243624.3.0000.5505
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis Knee; Chronic Pain
Keywords: Knee Osteoarthritis; Chronic Pain; Denervation; Radiofrequency Ablation; Chemical Neurolysis; Alcohol Neurolysis; Genicular Nerve Ablation; Minimally Invasive Pain Management; Interventional Pain Treatment; Pain Relief
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Group A - Continuous Ablative Radiofrequency Group B - Chemical Denervation with Absolute Alcohol
Who Masked: Outcomes Assessor
Masking Description: This study will use single-blind masking, where participants will be unaware of which treatment they receive. The physicians performing the procedures will not be blinded due to the nature of the interventions. However, the outcome assessors and data analysts will be blinded to the treatment allocation to minimize bias in pain assessments, functional evaluations, and overall study results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous Ablative Radiofrequency (Active Comparator): Participants in this arm will undergo continuous ablative radiofrequency targeting the sensory genicular nerves responsible for knee pain. The procedure involves the percutaneous insertion of a radiofrequency probe near the targeted nerves under imaging guidance. Controlled thermal energy will be applied to create a lesion, disrupting pain signal transmission. The goal is to provide long-lasting pain relief and improve function in patients with knee osteoarthritis.
  Interventions: Procedure: Continuous Ablative Radiofrequency
- Chemical Denervation with Absolute Alcohol (Active Comparator): Participants in this arm will undergo chemical denervation with absolute alcohol, targeting the sensory genicular nerves responsible for knee pain. The procedure involves the percutaneous injection of absolute alcohol near the selected nerves under imaging guidance. The neurolytic effect of alcohol disrupts pain signal transmission, aiming to provide prolonged pain relief and functional improvement in patients with knee osteoarthritis.
  Interventions: Drug: Chemical Denervation with Absolute Alcohol

INTERVENTIONS:
Procedure: Continuous Ablative Radiofrequency — Continuous ablative radiofrequency is a minimally invasive neuroablative procedure that targets the sensory genicular nerves to manage pain in knee osteoarthritis. Under ultrasound guidance, a radiofrequency probe is inserted percutaneously near the target nerves. The procedure delivers continuous thermal energy at 80°C for 120 seconds, creating a controlled lesion that disrupts pain signal transmission. This technique is distinct from pulsed radiofrequency, as it aims for permanent nerve ablation rather than neuromodulation. The expected outcome is prolonged pain relief and improved function in patients with chronic knee osteoarthritis refractory to conservative treatments.
  Arms: Continuous Ablative Radiofrequency
Drug: Chemical Denervation with Absolute Alcohol — Chemical denervation with absolute alcohol is a minimally invasive neurolytic procedure targeting the sensory genicular nerves to manage chronic knee osteoarthritis pain. Under ultrasound guidance, a percutaneous injection of absolute alcohol 66% is administered near the targeted nerves. The neurolytic effect of alcohol induces axonal degeneration and Wallerian degeneration, leading to prolonged disruption of pain signal transmission. This intervention differs from radiofrequency ablation as it achieves chemical neurolysis rather than thermal ablation, with potential for a distinct duration of analgesia and varying nerve regeneration patterns. The expected outcome is long-lasting pain relief and improved function in patients with knee osteoarthritis who have not responded to conservative treatments.
  Arms: Chemical Denervation with Absolute Alcohol

SUMMARY:
This randomized clinical trial compares two minimally invasive treatments for knee osteoarthritis pain that has not responded to conventional therapies. The study evaluates the effectiveness and safety of continuous ablative radiofrequency, which uses heat energy to disrupt pain signals, and chemical denervation with absolute alcohol, which involves an injection to reduce pain transmission. Participants will be randomly assigned to one of the treatments, and their pain levels, mobility, and quality of life will be monitored over time to determine which method provides better pain relief.

DETAILED DESCRIPTION:
This randomized clinical trial compares continuous ablative radiofrequency and chemical denervation with absolute alcohol for pain relief in patients with knee osteoarthritis refractory to conventional treatments. Participants will be randomly assigned to one of the two procedures, with outcomes assessed based on pain reduction, functional improvement, quality of life, and safety. Follow-ups will be conducted for up to six months to evaluate the durability of pain relief, providing evidence to guide clinical management of chronic knee osteoarthritis pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years.
* Knee pain for more than 3 months.
* Clinical and imaging-confirmed diagnosis of knee osteoarthritis, based on X-ray, ultrasound, or magnetic resonance imaging (MRI).

Exclusion Criteria:

* History of major joint interventions, such as previous knee surgery or arthroplasty.
* Severe joint effusion.
* Coagulation disorders or other clinical contraindications for the procedure.
* Uncontrolled comorbidities that increase procedural risk.
* Body mass index (BMI) > 35.
* Cognitive impairment that affects the ability to understand and respond to pain assessment instruments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Score | 6 months
  a validated questionnaire used to assess pain, stiffness, and physical function in patients with knee osteoarthritis. It consists of 24 items divided into three subscales: pain (5 items), stiffness (2 items), and physical function (17 items). Each item is rated on a Likert scale (0-4), with higher scores indicating greater pain, stiffness, and functional impairment. The total WOMAC score will be measured at baseline, 1 month, 3 months, and 6 months post-intervention to evaluate the effectiveness of the treatments in improving knee osteoarthritis symptoms.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) for Pain | 6 months
  The Numerical Rating Scale (NRS) is an 11-point scale (0-10) used to assess pain intensity, where 0 indicates "no pain" and 10 indicates "worst pain imaginable." Participants will rate their pain at rest and during movement at baseline, 1 month, 3 months, and 6 months post-intervention. The NRS is a widely used and validated tool for quantifying pain perception, allowing for objective comparison of pain relief between continuous ablative radiofrequency and chemical denervation with absolute alcohol.
Short Form-36 Health Survey (SF-36) | 6 months
  The SF-36 (Short Form-36 Health Survey) is a validated questionnaire used to assess health-related quality of life (HRQoL) across eight domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional health, and mental health. Scores range from 0 to 100, with higher scores indicating better health status and quality of life. The SF-36 will be administered at baseline, 1 month, 3 months, and 6 months post-intervention to evaluate the impact of continuous ablative radiofrequency and chemical denervation with absolute alcohol on the overall well-being of patients with knee

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo - Hospital Sao Paulo,, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No